CLINICAL TRIAL: NCT00728728
Title: Pregnenolone for Cognitive and Negative Symptoms in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MHBB-012-07F; NCT00639886 (obsolete NCT alias)
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: pregnenolone; schizophrenia; cognitive; positive symptom; negative symptom; placebo control
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Pregnenolone (Active Comparator): Pregnenolone
  Interventions: Drug: Dietary Supplement: Pregnenolone
- Arm 2: Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Dietary Supplement: Pregnenolone — Pregnenolone 50mg BID x 14 days, followed by Pregnenolone 150 x 14 days, followed by Pregnenolone 250 mg BID x thereafter for the remainder of the 8-week trial.
  Arms: Arm 1: Pregnenolone
Dietary Supplement: Placebo — Placebo
  Arms: Arm 2: Placebo

SUMMARY:
This study will investigate adjunctive pregnenolone for patients with schizophrenia and schizoaffective disorder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: DSM-IV/DSM-IV TR schizophrenia or schizoaffective disorder;
* Gender: Males and Females;
* Age: 21-65;
* Caucasian or Non Caucasian;
* Capable of providing informed consent;
* Duration of illness equal to or greater than one year;
* No change in antipsychotic medication in the previous eight weeks, no change in antipsychotic dose in the previous four weeks;
* No benzodiazepine use in the past twelve hours prior to cognitive testing;
* The patient cohort will be enriched for cognitive symptoms (Composite BACS scores = 0-3 standard deviations below the mean, assessed at the screening visit).

Exclusion Criteria:

* Subjects with a DSM-IV/DSM-IV TR diagnosis of alcohol or substance dependence (other than nicotine) within the last month;
* Subjects with a history of significant head injury/trauma, as defined by one or more of the following:

  * Loss of consciousness (LOC) for more than 1 hour,
  * Recurring seizures resulting from the head injury,
  * Clear cognitive sequelae of the injury,
  * Cognitive rehabilitation following the injury;
* Subjects with unstable medical illness or neurological illness (seizures, CVA);
* Patients with hormone-sensitive tumors (such as breast, uterine, or prostate cancer);
* Clinically significant abnormalities in physical examination , ECG, or laboratory assessments;
* Pregnant women or women of child-bearing potential, who are either not surgically-sterile or not using appropriate methods of birth control (serum beta-human chorionic gonadotropin [HCG] will be performed at baseline, 4 weeks, and 8 weeks to exclude pregnancy);
* Women who are breast-feeding;
* Electroconvulsive therapy (ECT) treatment within the last 3 months;
* Use of oral contraceptives or other hormonal supplementation such as estrogen. Although early studies suggested no effects on menstrual cycle, alterations in downstream metabolites of pregnenolone (such as estradiol) could theoretically impact the efficacy of oral contraceptives and/or estrogen replacement. Similarly, it is theoretically possible that pregnenolone could be metabolized to other steroids, resulting in hair, skin, or other steroid-related changes. Since we have determined in our prior study that pregnenolone administration does not result in downstream elevations in DHEA, DHEAS, estradiol, or testosterone, these possibilities may be unlikely;
* Current active suicidal and/or homicidal ideation, intent, or plan;
* Known allergy to study medication.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-12; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Marx, MD MA, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 2: Placebo: Placebo control group
Period: Overall Study
Arm/Group | Arm 1: Pregnenolone | Arm 2: Placebo
Started | 42 | 46
Completed | 38 | 34
Not Completed | 4 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Pregnenolone | Arm 2: Placebo | Total
Number analyzed (Participants) | 42 | 46 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (8.5) | 51.6 (8.4) | 51.7 (8.4)
Gender [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 36 | 39 | 75
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 36 | 63
  White | 12 | 9 | 21
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 46 | 88

OUTCOME MEASURES:

1. Primary Outcome: MATRICS Consensus Cognitive Battery (MCCB)
Description: The MATRICS Consensus Cognitive Battery (MCCB) is a standardized battery for use with adults with schizophrenia and related disorders to measure cognition in these individuals. The MCCB consists of ten individually administered test which measure speed of processing, attention/vigilance, nonverbal working memory, verbal working memory, verbal learning, visual learning, reasoning and problem solving and social cognition.
  The primary raw scores are entered into the MCCB Computer Scoring Program which then generates the corresponding T-scores and percentiles, along with a graphic profile of the scores for each of the seven cognitive domains. Higher scores indicate better performance.
Time Frame: Prospective, outcome measures collected over 10 week trial period. (Weeks 2, 6 and 10)
Measure: Mean (Standard Error); unit: T score
Arm/Group | Arm 1: Pregnenolone | Arm 2: Placebo
Number analyzed (Participants) | 38 | 34
T score
  Baseline | 30.92 (1.83) | 30.32 (1.40)
  Week 4 | 33.43 (1.75) | 32.76 (1.72)
  Week 8 | 36.97 (1.90) | 34.25 (2.11)

2. Primary Outcome: University of California Performance-based Skills Assessment (UPSA)
Description: The UCSD Performance-based Skills Assessment (UPSA) is a measure of Functional Capacity and assesses skills involved in community tasks. It is composed of five subdomains (comprehension and planning, finance, communication, mobility and house management) when combined, measures functional capacity. The comprehension and planning subdomain ranges from 0 to 14, the finance subdomain ranges from 0 to 11, the communication subdomain ranges from 0 to 12, the mobility subdomain ranges from 0 to 9, and the house management subdomain ranges from 0 to 4. Then a medication management score of 0 to 37 is added. In total, the Assessment is thus scored on a 0 to 87 scale, with higher scores indicating better performance.
Time Frame: Prospective, outcome measures collected over 10 week trial period. (Weeks 2, 6 and 10)
Measure: Mean (Standard Error); unit: total score
Arm/Group | Arm 1: Pregnenolone | Arm 2: Placebo
Number analyzed (Participants) | 38 | 34
total score
  Baseline | 77.49 (1.63) | 76.68 (1.76)
  Week 4 | 77.29 (2.65) | 80.12 (1.63)
  Week 8 | 85.63 (1.31) | 82.03 (2.05)

3. Primary Outcome: Brief Assessment of Cognition in Schizophrenia (BACS)
Description: The Brief Assessment of Cognition in Schizophrenia (BACS) captures those domains of cognition that are the most severely affected in patients with schizophrenia and the most strongly correlated with functional outcome. The domains of cognitive function assessed and the associated tests include: Verbal Memory & Learning (Verbal Memory), Working Memory (Digit Sequencing), Motor Function (Token Motor Task), Verbal Fluency (Semantic and Letter Fluency), Speed of Processing (Symbol Coding), and Executive Function (Tower of London). These domains are then converted to Z scores compared to standardized scoring scales, with higher scores representing better performance.
Time Frame: Prospective, outcome measures collected over 10 week trial period. (Weeks 2, 6 and 10)
Measure: Mean (Standard Error); unit: Z score
Arm/Group | Arm 1: Pregnenolone | Arm 2: Placebo
Number analyzed (Participants) | 38 | 34
Z score
  Baseline | -1.37 (0.13) | -1.53 (0.12)
  Week 4 | -1.11 (0.14) | -1.17 (0.12)
  Week 8 | -0.79 (0.13) | -1.09 (0.18)

4. Primary Outcome: Scale for the Assessment of Negative Symptoms(SANS)
Description: The Scale for the Assessment of Negative Symptoms (SANS) is an assessment used to obtain clinical ratings of negative symptoms in patients with schizophrenia. The SANS assesses five symptom complexes. They are: affective blunting; alogia (impoverished thinking); avolition/apathy; anhedonia/asociality; and disturbance of attention. 24 assessments are conducted on a six-point scale (0=not at all to 5=severe) each, for a total scoring range of 0-120. Lower scores represent better performance.
Time Frame: Prospective, outcome measures collected over 10 week trial period. (Weeks 2, 6 and 10)
Measure: Mean (Standard Error); unit: total score
Arm/Group | Arm 1: Pregnenolone | Arm 2: Placebo
Number analyzed (Participants) | 38 | 34
total score
  Baseline | 26.92 (1.75) | 25.88 (1.94)
  Week 4 | 23.87 (2.05) | 21.74 (1.87)
  Week 8 | 21.00 (2.47) | 20.77 (2.40)

5. Secondary Outcome: The Calgary Depression Scale for Schizophrenia (CDSS)
Description: The CDSS assesses the level of depression in schizophrenia by measuring nine items on a 0 (absent) to 3 (severe) scale each. Thus, the total score range is 0 to 27. Lower scores represent better outcomes.
Time Frame: Prospective, outcome measures collected over 10 week trial period.
Measure: Mean (Standard Error); unit: total score
Arm/Group | Arm 1: Pregnenolone | Arm 2: Placebo
Number analyzed (Participants) | 38 | 34
total score
  Baseline | 2.84 (0.64) | 3.18 (0.64)
  Week 4 | 2.39 (0.62) | 2.79 (0.66)
  Week 8 | 2.68 (0.74) | 2.46 (0.90)

6. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: The PANSS measures positive and negative symptoms of schizophrenia through administering a structured interview. After the interview, 25 PANSS items are each rated 1 (absent) to 7 (extreme). These items are organized into five scales: Negative, Positive, Dysphoric Mood, Activation, and Autistic Preoccupation. The combination of the 25 items produces a total score range of 25-175, and lower scores represent better outcomes.
Time Frame: Prospective, outcome measures collected over 10 week trial period. (Weeks 2, 6 and 10)
Measure: Mean (Standard Error); unit: total score
Arm/Group | Arm 1: Pregnenolone | Arm 2: Placebo
Number analyzed (Participants) | 38 | 34
total score
  Baseline | 65.74 (2.28) | 63.68 (2.58)
  Week 4 | 61.47 (2.55) | 56.79 (2.03)
  Week 8 | 59.10 (2.95) | 57.12 (3.16)

7. Secondary Outcome: Clinical Global Impressions (CGI) Scale
Description: The CGI scale provides a brief, stand-alone assessment of the clinician's view of the patient's global functioning prior to and after initiating a study medication. The CGI comprises two companion one-item measures evaluating the severity of psychopathology from 1 to 7 and change from the initiation of treatment on a similar seven-point scale. Thus, scores range from 2 to 14, with lower scores representing better outcomes.
Time Frame: Prospective, outcome measures collected over 10 week trial period. (Weeks 2, 6 and 10)
Population: Missing data for a total of 5 participants for the CGI.
Measure: Mean (Standard Error); unit: score
Arm/Group | Arm 1: Pregnenolone | Arm 2: Placebo
Number analyzed (Participants) | 34 | 33
score
  Baseline | 3.56 (0.15) | 3.58 (0.13)
  Week 4 | 3.39 (0.12) | 3.39 (0.14)
  Week 8 | 3.42 (0.12) | 3.24 (0.17)

ADVERSE EVENTS:
Arm/Group | Arm 1: Pregnenolone | Arm 2: Placebo
Serious Adverse Events (participants affected / at risk) | 3/42 | 4/46
Other Adverse Events (participants affected / at risk) | 31/42 | 38/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Pregnenolone (N=42) | Arm 2: Placebo (N=46)
Psychiatric Hopitalization (Psychiatric disorders) | 2 | 2
Hospitalization for Elevated Glucose (Endocrine disorders) | 1 | 0
Medical Admission for Observation (Gastrointestinal disorders) | 0 | 1
Breast Cancer Diagnosis (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Pregnenolone (N=42) | Arm 2: Placebo (N=46)
Drowsiness (Nervous system disorders) | 11 | 10
Hypersomnia (Nervous system disorders) | 9 | 8
Diarrhea (Gastrointestinal disorders) | 8 | 7
Insomnia (Nervous system disorders) | 7 | 3
Decreased Appetite (Nervous system disorders) | 8 | 6
Increased appetite (Nervous system disorders) | 7 | 9
Constipation (Gastrointestinal disorders) | 5 | 12
Nausea (Gastrointestinal disorders) | 6 | 2
Dry mouth (Nervous system disorders) | 5 | 8
Cramps (Musculoskeletal and connective tissue disorders) | 7 | 6
Headache (Nervous system disorders) | 6 | 9
Tremor (Nervous system disorders) | 5 | 5
Increased Salivation (Nervous system disorders) | 5 | 1
Palpitations (Cardiac disorders) | 4 | 7
Tinnitus (Ear and labyrinth disorders) | 3 | 5
Dermatological (Skin and subcutaneous tissue disorders) | 3 | 4
Joint pain/ stiffness (Musculoskeletal and connective tissue disorders) | 5 | 2
Dizziness (Nervous system disorders) | 4 | 9
Sweating (Nervous system disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Muscle Pain/Stiffness (Musculoskeletal and connective tissue disorders) | 3 | 4
Other: "Lucid Dreams" (Nervous system disorders) | 1 | 0
Restlessness (General disorders) | 3 | 4
Nocturnal/Enuresis (Renal and urinary disorders) | 1 | 1
Decreased Interest in Sex (Nervous system disorders) | 2 | 0
Vertigo (Nervous system disorders) | 1 | 0
Blurred Vision (Eye disorders) | 1 | 4
Menstrual Disturbance (Reproductive system and breast disorders) | 1 | 0
Nasal Congestion (General disorders) | 1 | 4
Peripheral Edema (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 1
Akathisia (Musculoskeletal and connective tissue disorders) | 1 | 0
Excitement/Agitation (Nervous system disorders) | 1 | 1
Confusion (Nervous system disorders) | 1 | 2
Paresthesia (Nervous system disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 1
Increased Motor Activity (Musculoskeletal and connective tissue disorders) | 0 | 1
Cold Extremities (Blood and lymphatic system disorders) | 0 | 1
Other: "Urinary Retention" (Renal and urinary disorders) | 0 | 1
Other: "Head/Neck Twitching" (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes